CLINICAL TRIAL: NCT04198116
Title: Combining Varenicline and Guanfacine for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sherry McKee, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000026630; R01DA047986 (NIH)
Record Dates: First submitted 2019-12-03; First posted 2019-12-13 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline; Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Varenicline + Guanfacine ER (Experimental): Varenicline (2mg/day) + Guanfacine extended release (6mg/day ER). Varenicline (2mg/day) administered orally twice a day at 8:00 AM and 8:00 PM while titrating to full dose. Titration schedule: Days 1-9 0mg/day; 0mg/dose, Days 10-12 0.5mg/day; 0.5mg/dose 8:00 PM, Days 13-15 1mg/day; 0.5mg/dose, Days 16-21 2mg/day; 1mg/dose. Guanfacine ER (6mg/day) administered orally twice daily at 8:00 AM and 8:00 PM while titrating to the full dose. Titration schedule: Days 1-3 1mg/day; 0.5mg/dose, Days 4-6 2mg/day; 1mg/dose, Days 7-9 3mg/day; 1.5mg/dose, Days 10-12 4mg/day; 2mg/dose; Days 13-15 5mg/day; 2.5mg/dose and Days 16-23 6mg/day; 3mg/dose. Once at steady state, administration is orally once per day at 8:00 PM for both medications.
  Interventions: Drug: Varenicline; Drug: Guanfacine ER
- Varenicline (Active Comparator): Varenicline (2mg/day). Varenicline (2mg/day) administered orally twice a day at 8:00 AM and 8:00 PM while titrating to full dose. Titration schedule: Days 1-9 0mg/day; 0mg/dose, Days 10-12 0.5mg/day; 0.5mg/dose 8:00 PM, Days 13-15 1mg/day; 0.5mg/dose, Days 16-21 2mg/day; 1mg/dose. Once at steady state, administration is orally once per day at 8:00 PM.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline 2mg/day
  Other Names: Chantix
Drug: Guanfacine ER — Guanfacine Extended Release (6mg/day ER)
  Other Names: Intuniv
  Arms: Varenicline + Guanfacine ER

SUMMARY:
The novel design of this study combines a laboratory paradigm to evaluate stress-induced smoking behavior and smoking-related reinforcement, followed by a 12-week treatment phase to evaluate clinical outcomes.

DETAILED DESCRIPTION:
Using a double-blind, this Phase 2 study will randomize 140 smokers to a parallel group design (varenicline + guanfacine vs. varenicline alone). Following titration to steady state levels, the investigators will evaluate sex differences in medication effects on stress-induced smoking behavior and smoking-related reinforcement in the laboratory, and on abstinence outcomes during a subsequent 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. Able to read and write English
3. SMOKER: 10 or more cigarettes per day for at least the past year, Carbon Monoxide (CO) > 10 ppm at intake
4. Able to take oral medications and willing to adhere to medication regimen
5. Provide evidence of a stable living residence in the last 2 months prior to randomization, have reasonable transportation arrangements to the study site, have no plans to move within the next 3 months, and have no unresolved legal problems
6. Motivated to quit smoking (8 or greater on the Contemplation Ladder)

Exclusion Criteria:

1. Subjects with any significant current medical conditions (neurological, cardiovascular [including hypertension or hypotension: sitting BP >160/100 or <90/60mmHg at baseline screening], endocrine, thyroid, renal, liver), seizures, delirium or hallucinations, or other unstable medical conditions
2. Current Diagnostic and Statistical Manual of Mental Disorders (DSM-V) alcohol or substances use disorders, other than mild alcohol use disorder or tobacco use disorder
3. Subjects who have a positive test result at intake appointment on urine drug screens conducted for illicit drugs
4. Past 30 day use of psychoactive drugs excluding anxiolytics and antidepressants (however, see #10; barbiturates, benzodiazepines are exclusionary)
5. Women who are pregnant or nursing, or fail to use one of the following methods of birth control unless she or partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or IUD)
6. Suicidal, homicidal or evidence of current (past 6-month) severe mental illness such as schizophrenia or bipolar disorder
7. meeting DSM-V criteria for current (past-6 month) attention deficit hyperactivity disorder (ADHD)
8. Individuals who are currently taking medications known to be effective for smoking cessation (e.g., FDA smoking cessation medications, nortriptyline, clonidine) or are regular users of e-cigarettes or other tobacco projects (pipe, cigar, smokeless tobacco) in the past 30 days
9. Only one member per household can participate in the study
10. Specific exclusions for administration of guanfacine not already specified: EKG evidence at baseline screening of any clinically significant conduction abnormalities or arrhythmias; known intolerance for guanfacine or any alpha blocker; history of fainting, syncopal attacks, heart failure or myocardial infarction, or impaired liver (aspartate aminotransferase [AST], alanine aminotransferase [ALT] > 3x normal) or renal function (estimated creatinine clearance <60 cc/min); treatment with any antihypertensive drug or any alpha-blocker; use of any central nervous system (CNS) depressant (e.g., phenothiazines, barbiturates, benzodiazepines)
11. Specific exclusions for the administration of varenicline not already specified: known intolerance to varenicline or taking H2blockers (e.g., Cimetidine), quinolones, or trimethoprim.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Latency | 50 minutes
  Latency (in minutes) to time of first cigarette smoked during the delay period.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No